CLINICAL TRIAL: NCT00489190
Title: Local, Open, Non-Randomized, Phase IV Clinical Study for the Collection of Data Regarding the Drug Portability Received During the Treatment With Subcutaneous Injection of Apidra Glulisine (HMR1964) to Patients With Diabetes Mellitus 1st Type
Brief Title: APIDRA Registration Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APIDR_L_00041
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine

INTERVENTIONS:
Drug: Insulin Glulisine

SUMMARY:
To collect effectiveness and safety data during the treatment with Apidra glulisine (HMR1964) by means of subcutaneous injections to patients with Diabetes Mellitus 1st type during 12 weeks-active phase.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus 1st type, with НbA1c level in the range of ≥ 6,5 - <=11%, receiving the regimen of multiple injections of insulin during one year.

Exclusion Criteria:

* Active proliferative diabetic retinopathy connected with focal or panretinal photocoagulation or vitrectomy carried out within 6 months before visit 1, or any unstable (quickly progressive) form of retinopathy, which may need in surgical intervention (including laser photocoagulation) during study
* Diabetes Mellitus of the 2nd type
* Patients transmitted pancreatectomy
* Patients transmitted transplantation of pancreas or islet cells
* Probable therapy by means of products not approved by study minutes during the study
* Anamnestic indications of convulsive disorders
* Allergic reaction on insulin or any filler of preparation Apidra (glulisine)
* Clinical serious diseases of cardiovascular system, liver, nervous system, endocrine system, oncologic diseases or other serious system diseases, which complicate keeping of minutes or interpretation of study results, and, at the investigator's opinion, impede the safe participation of patients in study
* Drug addiction or alcoholism
* Disturbance of liver functions confirmed with the increase of ALT or AST activity up to the level twice as high as the upper standard limit (these indications may not be single)
* Disturbance of functions of kidneys confirmed with the level of creatinine in serum that is more than 177 mµmol/l at visit 1 (this indication may not be single)
* Pregnancy or breast-feeding

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-08

PRIMARY OUTCOMES:
Dynamics НbA1c in the final point compared with the initial level. | end of the study
Dynamics compared with the initial level of glycemia and insulin dosages. | 12 weeks

SECONDARY OUTCOMES:
Evaluation of frequency of glycemia episodes. Also undesirable events, Influence on indexes of general clinical analysis of blood and biochemical analysis of blood. | from the beginning to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Arman UTEGULOV, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Almaty, Kazakhstan